CLINICAL TRIAL: NCT01512914
Title: Impact of Intraperitonael Nebulization of Local Anesthetic on Postoperative Pain Associated With Laparoscopic Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: San Gerardo Hospital (Other)
Responsible Party: Principal Investigator, Pablo Mauricio Ingelmo M.D., MD, San Gerardo Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR HSG 01-2008
Record Dates: First submitted 2012-01-15; First posted 2012-01-19 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Gynecologic Laparoscopic Surgery
Keywords: Gynecologic laparoscopic surgery; Postoperative pain; Nebulization; Ropivacaine
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- CONTROL group (Placebo Comparator)
  Interventions: Drug: saline
- PREOPERATIVE nebulization (Experimental)
  Interventions: Drug: Ropivacaine 30 mg
- POSTOPERATIVE nebulization (Experimental)
  Interventions: Drug: Ropivacaine 30 mg
- INSTILLATION group (Active Comparator)
  Interventions: Drug: Ropivacaine 100 mg

INTERVENTIONS:
Drug: Ropivacaine 30 mg — preoperative instillation of saline 20 ml, nebulization of ropivacaine 1% 3 ml (30 mg) before surgery and nebulization of saline 3 ml after surgery
  Arms: PREOPERATIVE nebulization
Drug: Ropivacaine 30 mg — preoperative instillation of saline 20 ml, preoperative nebulization of saline 3 ml and nebulization of ropivacaine 1% 3 ml (30 mg) after surgery
  Arms: POSTOPERATIVE nebulization
Drug: Ropivacaine 100 mg — preoperative instillation of ropivacaine 0,5% 20 ml (100 mg) and nebulization of saline 3 ml before and after surgery
  Arms: INSTILLATION group
Drug: saline — preoperative instillation of saline 20 ml and nebulization of saline before and after surgery
  Arms: CONTROL group

SUMMARY:
Studies evaluating intraperitoneal local anesthetic instillation for pain relief after laparoscopic procedures have provided conflicting results. This randomized, double-blind study was designed to assess the effects of a novel intraperitoneal local anesthetic administration technique using nebulization on pain relief after gynecologic laparoscopic surgery.

DETAILED DESCRIPTION:
Studies evaluating intraperitoneal local anesthetic (LA) instillation for pain relief after laparoscopic surgery have provided conflicting results. One of the factors that might contribute to failure of the instillation technique may be related to inadequate distribution of local anesthetic throughout the peritoneal surface. In contrast, nebulization should provide a uniform spread of drugs throughout the peritoneal cavity and thus may be beneficial to improve pain relief after laparoscopic procedures. The investigators reported that a microvibration-based nebulization device (Aeroneb Pro® system, Aerogen, Galway, Ireland) could be used for ropivacaine delivery into the insufflation gas required to create pneumorpeitoneum. The investigators hypothesized that intraperitoneal ropivacaine nebulization would provide superior pain relief than ropivacaine instillation after gynecologic laparoscopic surgery. This randomized, double blind, controlled clinical trial was designed to assess the analgesic efficacy of ropivacaine nebulization before or after surgery compared with intraperitoneal ropivacaine instillation and placebo after gynecologic laparoscopic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Females 18-70 years old, ASA score 1 - 3;
* scheduled for laparoscopic operative surgery in the Obstetrics and Gynecology unit;
* free from pain in preoperative period, without habitual analgesic use;
* without cognitive impairment or mental retardation, who gave a written informed consent

Exclusion Criteria:

* Females under 18 or over 70;
* ASA 4 or 5;
* emergency/urgency criteria, postoperative admission in a intensive care unit with sedation or ventilatory assistance; cognitive impairment or mental retardation;
* habitual analgesic use; progressive degenerative diseases of the CNS;
* convulsions or chronic therapy with antiepileptic drugs;
* severe hepatic or renal impairment;
* pregnancy or lactation;
* allergy to one of the specific substances used in the study;
* acute infectious disease or inflammatory chronic disease, alcohol or drug addiction;
* any kind of communication problem;
* neurologic or psychiatric disease;
* no written informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
postoperative pain | 24 hours
  Postoperative pain was assessed by NRS (0 to 10 points) at rest (static NRS) and after a deep inspiration or cough (dynamic NRS). The proportion of patients with adequate pain control after surgery (dynamic NRS < 3) will also be assessed.

SECONDARY OUTCOMES:
morphine consumption | 24 hours
  The total dose of morphine at every evaluation after awakening will be quantified using the PACU clinical chart and/or PCA infusers memory display
Unassisted walking time | 24 hours
  Unassisted walking time is defined as the time in hours between PACU discharge and when the patient is able to walk out of his room and back to bed without any assistance.
Hospital stay | between surgery and discharge
  We define hospital stay as the elapsed time between surgery and hospital discharge
hospital morbidity | up to discharge
  All complications or adverse effects associated or possibly associated with the interventions under study, surgery or anesthesia will be quantified using the anesthesia charts, surgical charts, surgical database.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo M Ingelmo, MD, Principal Investigator — San Gerardo Hospital
Locations (1):
- San Gerardo Hospital, Monza, MB, Italy

REFERENCES:
- [Result] Goldstein A, Grimault P, Henique A, Keller M, Fortin A, Darai E. Preventing postoperative pain by local anesthetic instillation after laparoscopic gynecologic surgery: a placebo-controlled comparison of bupivacaine and ropivacaine. Anesth Analg. 2000 Aug;91(2):403-7. doi: 10.1097/00000539-200008000-00032. PMID 10910857
- [Result] Alkhamesi NA, Peck DH, Lomax D, Darzi AW. Intraperitoneal aerosolization of bupivacaine reduces postoperative pain in laparoscopic surgery: a randomized prospective controlled double-blinded clinical trial. Surg Endosc. 2007 Apr;21(4):602-6. doi: 10.1007/s00464-006-9087-6. Epub 2006 Dec 16. PMID 17180268
- [Result] Greib N, Schlotterbeck H, Dow WA, Joshi GP, Geny B, Diemunsch PA. An evaluation of gas humidifying devices as a means of intraperitoneal local anesthetic administration for laparoscopic surgery. Anesth Analg. 2008 Aug;107(2):549-51. doi: 10.1213/ane.0b013e318176fa1c. PMID 18633034